CLINICAL TRIAL: NCT06993831
Title: ENGAGE Pilot Study: Alleviating Negative Symptoms in Schizophrenia Using a Virtual Reality-based Intervention Targeting Social Reward Learning
Brief Title: ENGAGE: Virtual Reality-based Psychotherapy for Negative Symptoms in Schizophrenia
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24046055; H-24046055 (Other: De Videnskabsetiske Komiteer for Region Hovedstaden)
Record Dates: First submitted 2025-02-21; First posted 2025-05-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia Spectrum Disorders; Negative Symptoms in Schizophrenia
Keywords: schizophrenia; psychotherapy; VR; psychosocial intervention; psychosis; negative symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — engage 8200

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Participants randomized to this arm will not receive any treatment beyond the standard care offered by the usual health care providers.
- VR-based psychotherapy (Experimental): Participants randomized to this arm will receive 10 sessions of the VR-based intervention targeting negative symptoms in schizophrenia in addition to any possible treatment offered by other health care providers.
  Interventions: Behavioral: Virtual Reality-based psychotherapy

INTERVENTIONS:
Behavioral: Virtual Reality-based psychotherapy — A manualized, modularized, Virtual Reality-based intervention comprising 10 sessions of 1 hour each. The VR therapy aims at enhancing anticipatory pleasure and positive emotions by amplifying exposure and reactivity towards social environments and rewarding activities using a highly elaborate VR software. The VR exposure comprises several different virtual social environments (e.g., a bus, a café, a park etc.) In a tailored treatment approach, therapists will guide participants to train focusing on positive stimuli, engage in activities, experience social rewards, and practice expressing emotions through body language.
  The therapy focuses on increasing the awareness of positive outcomes that may influence motivation. The therapy deploys activity appraisal/re-appraisal intended to enhance the salience of future opportunities for reward and desire for such rewards, thus targeting reward anticipation processes and promoting enjoyable daily-life activities.
  Other Names: ENGAGE
  Arms: VR-based psychotherapy

SUMMARY:
The primary goal of this pilot study is to examine the feasibility and acceptability of a new Virtual Reality-based intervention against negative symptoms in schizophrenia spectrum disorders (SSD).

The main questions it aims to answer are:

1. Is Virtual Reality-based therapy a feasible and acceptable treatment for negative symptoms in SSD?
2. Are there indications that the treatment is effective in reducing negative symptoms, improving daily functioning, and enhancing quality of life?

Researchers will compare the new Virtual Reality-based treatment to standard psychiatric care to evaluate therapy effectiveness.

Participants will be allocated to receive either 10 sessions of Virtual Reality-based therapy or Treatment as usual. All participants will undergo a thorough assessment at baseline and at follow-up after 12 weeks.

DETAILED DESCRIPTION:
Negative symptoms (NS) are core features of schizophrenia and strongly correlated with vocational and social outcomes, quality of life, and have a higher impact on later outcome than positive symptoms (PS) such as hallucinations and delusions. While there are good medical treatment options for PS, no robust and replicated evidence exists for effective NS treatments. Consistent evidence suggests that abnormalities of the brain reward system are central in the pathogenesis of NS, i.e., the domains of anhedonia and avolition. Preliminary evidence indicates changes in reward learning following therapy is related to a reduction in NS.

Virtual reality (VR) is a promising technologically advanced mental health research tool with high ecological validity. VR allows individuals to immerse themselves in realistic environments and interact with virtual objects, providing a safe and controlled space to address symptoms and improve functioning. Initial evidence (N=4) supports that VR-based interventions significantly reduce NS and improve psychosocial functioning with a medium to large effect size. Given the suggested central role of reward processing disturbances in the pathogenesis of NS, there is an obvious need to investigate the effect of a VR-based intervention targeting reward processing in ameliorating NS.

Both NS and motivational abnormalities reflect complex processes at a system level likely corresponding to functional brain activity within and between several regions and circuits. Supplementing the clinical assessments in the study with magnetic resonance imaging (MRI) data may clarify whether the intervention directly targeting reward processing has an effect on the biological processes/networks involved.

In sum, this study will explore the prospects of using an innovative, VR-based treatment to treat NS and reward processing deficits in schizophrenia aimed at producing real-life benefits for the patients. If found successful, this pilot study could lay the foundation for a larger randomized clinical trial examining the intervention's effectiveness. Prospectively, these results can pave the way for a much sought-after treatment option for NS.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of a schizophrenia-spectrum disorder (F2x)
* Negative symptom score of ≥3 on the SANS items avolition or anhedonia

Exclusion Criteria:

* Diagnosis of organic brain disease
* Intellectual disability (IQ < 70)
* Current diagnosis of drug dependency
* Command of spoken Danish or English inadequate for engaging in therapy
* Refusing to be informed on incidental findings on the MRI scans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability as assessed by recruitment rate | Recruitment rate is monitored throughout the study period (15 months)
  Percentage of target sample (30 participants) recruited after 15 months from study start
Feasibility and acceptibility as assessed by retention rate | Retention rates are monitored throughout the study period (15 months)
  Percentage of included participants in the experimental group who retent to treatment at cessation of therapy (10 sessions)
Feasibility and acceptability as assessed by level of satisfaction in the experimental group | At 12 weeks follow-up
  Percentage of participants in the experimental group reporting a satisfaction rating of more than 7 on a 10-point Likert scale with higher scoring indicating a higher level of satisfaction with therapy.

SECONDARY OUTCOMES:
Severity of negative symptoms as assessed by the Brief Negative Symptoms Scale (BNSS) | Baseline and at 12 weeks follow-up
  The BNSS is a an interviewer-administered instrument comprising 13 items and five domains of negative symptoms: anhedonia, asociality, avolition, blunted effect and alogia.
  Each item is rated on a 7-point scale (0-6) with higher scores reflecting a higher level of negative symptoms.
Severity of negative symptoms as assessed by the Scale for the Assessment of Negative Symptoms (SANS) | Baseline and at 12 weeks follow-up
  The SANS is an interviewer-administered instrument comprising 23 items and four domains of negative symptoms: affective flattening or blunting, alogia, avolition-apathy, and anhedonia-asociality.
  Each item is rated on a 5-point scale (0-5) with higher scores reflecting a higher level of negative symptoms.
Severity of negative symptoms as assessed by the Self-evaluation of Negative Symptoms (SNS) | Baseline and at 12 weeks follow-up
  The SNS is a patient questionnaire comprising 20 items and 5 domains of negative symptoms: social withdrawal, diminished emotional range, alogia, avolition, and anhedonia.
  Each item is rated on a 3-point scale (0-2) with higher scores reflecting higher levels of negative symptoms.
Social and daily functioning as assessed by the Personal and Social Performance Scale (PSP) | Baseline and at 12 weeks follow-up
  The PSP is an interviewer-administered instrument assessing different domains of social and daily functioning: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior.
  A score between 1-100 is assigned with higher scores indicating better functioning.
Social functioning as assessed by the Social Functioning Scale (SFS) | Baseline and at 12 weeks follow-up
  The SFS is a self-report instrument assessing social functioning among individuals with schizophrenia.
  The instrument comprises seven domains: Social engagement/withdrawal, Interpersonal behaviour, Prosocial activities, Recreation, Independence-competence, Independence-performance and Employment/occupation.
  The minimum raw score is 0 and maximum raw score is 223 with higher scoring indicating a higher level of functioning.

OTHER OUTCOMES:
Psychological well-being as assessed by The World Health Organisation- Five Well-Being Index (WHO-5) | Baseline and at 12 weeks follow-up
  The WHO-5 is a self-report questionnaire with 5 items measuring subjective psychological well-being. Each item is scored on a 6-point scale ranging At no time (0) to All of the time (5).
  A total raw score is ranging from 0 to 25. To calculate the final score, the total raw score is multiplied by 4 with higher scores reflecting higher levels of well-being.
Level of depressive symptoms as assessed by the Calgary Depression Scale for Schizophrenia (CDSS) | Baseline and at 12 weeks follow-up
  The CDSS is an interviewer-administered instrument comprising 9 items assessing level of depression among individuals with schizophrenia. Each item is rated on a 4-point scale ranging from Absent (0) to Severe (3) with higher scores indicating a higher level of depressive symptoms.
Perceived interpersonal pleasure as assessed by the Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | Baseline and at 12 weeks follow-up
  The ACIPS is a patient questionnaire comprising 17 items assessing hedonic capacity for social interaction and interpersonal engagement.
  Each item is rated on a 6-point scale (1-6) with higher scores reflecting higher levels of hedonic capacity.
Defeatist performance beliefs as assessed by the Defeatist Performance Attitude Scale (DPAS) | Baseline and at 12 weeks follow-up
  The DPAS is a self-report instrument comprising 15 items assessing defeatist performance beliefs.
  Each item is rated on a 7-point scale (1-7) with higher scores reflecting stronger defeatist performance beliefs (range: 15-105).
Severity of positive symptoms as assessed by the Scale for the Assessment of Positive Symptoms (SAPS) | Baseline and at 12 weeks follow-up
  SAPS is an interviewer-administered instrument with 34 items measuring severity of hallucinations, delusions, bizarre behavior and positive formal thought disorder.
  Each item is rated on a 6-point scale (0-5) with higher scores reflecting higher levels of positive symptoms.
Emotion processing capability as assessed by the Emotion Recognition Task (CANTAB ERT) | Baseline and at 12 weeks follow-up
  Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise).The outcome measures for ERT cover percentage and number correct or incorrect and overall response latencies, which can be looked at either across individual emotions or across all emotions at once.
Readiness for therapy as assessed by the Readiness for Therapy Questionnaire (RTQ) | Baseline and at 12 weeks follow-up
  RTQ is a 6-item self-report questionnaire measuring the participants positive attitude and preparedness to enter therapy for the purpose of resolving problems. Each item is scored on a 5-point Likert scale ranging from strongly disagree (0) to strongly agree (4). Item 2, 3 and 6 are reversed scored. A higher score indicates greater readiness for therapy.
Client satisfaction as assessed by the Client Satisfaction Questionnaire (CSQ) | Baseline and at 12 weeks follow-up
  CSQ is an 8 item self-report measuring client satisfaction with the intervention. All items are scored on a 4-point Likert scale ranging from bad (1) to excellent (4). Higher scores indicate higher satisfaction.
Virtual Reality simulation sickness as assessed by the Virtual Reality Simulation Sickness Questionnaire, Modified Danish Version (VRSSQ-MDV) | Baseline and at 12 weeks follow-up
  VRSSQ-MDV is a is a self-report questionnaire measuring virtual reality simulation sickness. The Modified Danish Version consists of 9 items rated on a 4-point Likert Scale ranging from 0 (not at all) to 3 (a lot). Higher scores reflect higher degree of virtual reality simulation sickness. The VRSSQ-MDV will be administered only to participants in the experimental group.
Immersion in VR as assessed by the Multimodal Presence Scale, Modified Shortened Danish Version (MPS-MSDV) | Baseline and at 12 weeks follow-up
  MPS-MSDV is a self-report questionnaire measuring presence in virtual reality. The modified, shortened Danish Version consists of 10 selected items scored on a 5-point Likert Scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Higher scores reflect higher degree of presence in Virtual Reality. The MPS-MSDV will be administered only to participants in the experimental group.
Reward system activation in mesocorticolimbic and fronto-striatal circuits as assessed by functional magnetic resonance imaging (MRI) | Baseline and at 12 weeks follow-up
  Brain activation during anticipation of monetary and social rewards will be examined using two functional paradigms, the Social Incentive Delay Task (SIDT) and the Monetary Incentive Delay Task (MIDT). Key regions of interest for the study include mesocorticolimbic and fronto-striatal circuits including ventral tegmental area, amygdala, hippocampus, striatum, nucleus accumbens, and prefrontal cortex. Additionally, resting state fMRI will be acquired.
Positive affect (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints per day over a 7-day course. Using a purpose-designed questionnaire, positive affect will be measured on a 4-item visual analogue scale from 0 to 10 with higher values indicating greater positive affect.
Negative affect (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints per day over a 7-day course. Using a purpose-designed questionnaire, negative affect will be measured on a 4-item visual analogue scale from 0 to 10 with higher values indicating greater negative affect.
Consummatory and anticipatory hedonia (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints per day over a 7-day course. Using a purpose-designed questionnaire, consummatory and anticipatory hedonia in reaction to activities will be measured on a 2-item visual analogue scale from 0 to 10 with higher values indicating greater negative affect.
Number of self-reported activities (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints (beeps) per day over a 7-day course. Using a purpose-designed questionnaire, the number of self-reported activities at each beep and the number of beeps without any activities will be recorded.
Number of self-reported companions (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints (beeps) per day over a 7-day course. Using a purpose-designed questionnaire, the number of self-reported companions and the number of beeps in absence of company will be recorded.
Asociality (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints per day over a 7-day course. Using a purpose-designed questionnaire, asociality in reaction to being alone or in company will be measured on a 4-item visual analogue scale from 0 to 10 (of which two items are inversely coded) with higher values indicating greater asociality.
Avolition (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints per day over a 7-day course. Using a purpose-designed questionnaire, avolition will be measured on a 2-item visual analogue scale from 0 to 10 with lower values indicating greater levels of avolition.
Sedentary behavior (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints per day over a 7-day course. Time spent on sedentary behaviors will be calculated from accelerometry data recorded from participants' mobile phone sensors.
Time spent at home (Ecological Momentary Assessment) | Baseline and at 12 weeks follow-up
  Ecological Momentary Assessment (EMA) will be employed capturing momentary features of negative symptoms at 5 randomly distributed timepoints per day over a 7-day course. As an objectively measurable feature of inactivity, time spent at home will be calculated from location data recorded from participants' mobile phone sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Louise B Glenthøj, PhD, dr.med., Principal Investigator — VIRTU Research Group, Mental Health Center Copenhagen, Copenhagen University Hospital - Mental Health Services CPH, Denmark
Locations (1):
- Copenhagen Research Center for Mental Health (CORE), Mental Health Services CPH, Denmark, Hellerup, Greater Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donath VM, Ries ES, Mariegaard L, Kristensen TD, Ebdrup BH, Strauss GP, Fisher PM, Rostrup E, Nordentoft M, Hilker R, Melau M, Bockting CL, Albert N, van Bennekom MJ, Ambrosen KS, Glenthoj LB. Alleviating negative symptoms in schizophrenia using a virtual reality-based therapy targeting social reward learning (ENGAGE): Protocol for a randomised, controlled, assessor-blind pilot study. PLoS One. 2025 Oct 8;20(10):e0331632. doi: 10.1371/journal.pone.0331632. eCollection 2025. PMID 41060907